CLINICAL TRIAL: NCT05322200
Title: Potential Impact of Oral Semaglutide on Coronary Artery Disease Progression Following Acute Coronary Syndrome: The POST-ACS Study
Brief Title: The POST-ACS Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swansea Bay University Health Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 275165
Record Dates: First submitted 2022-02-11; First posted 2022-04-11 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus; Acute Coronary Syndrome; Coronary Artery Disease
MeSH Terms: conditions — Diabetes Mellitus; Acute Coronary Syndrome; Coronary Artery Disease | interventions — Hematologic Tests

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active drug (Active Comparator): Oral Semaglutide + conventional therapy (includes dual antiplatelets, Statin, Angiotensin-converting enzyme inhibitors (ACE inhibitors) and beta-blockers)
  Interventions: Radiation: A computerized tomography (CT) coronary angiogram; Procedure: Vicorder (Skidmore medical, UK); Other: Blood tests for inflammation and oxidative stress markers
- Placebo (Placebo Comparator): placebo (same dose and administration route) + conventional therapy (includes dual antiplatelets, Statin, Angiotensin-converting enzyme inhibitors (ACE inhibitors) and beta-blockers)
  Interventions: Radiation: A computerized tomography (CT) coronary angiogram; Procedure: Vicorder (Skidmore medical, UK); Other: Blood tests for inflammation and oxidative stress markers

INTERVENTIONS:
Radiation: A computerized tomography (CT) coronary angiogram — Participants in both arms will undergo CT coronary angiogram with Plaque Map analysis at baseline prior to therapy initiation and following 12 months of treatment.
Procedure: Vicorder (Skidmore medical, UK) — Participants in both arms will undergo aortic carotid-femoral pulse wave velocity (cfPWV)through the Vicorder (Skidmore medical, UK), which uses oscillometric cuff-based measurements to establish the index of arterial stiffness. The procedure will be done at baseline and 12 months after therapy initiation.
Other: Blood tests for inflammation and oxidative stress markers — All the participants will have (non-fasting) blood samples performed to assess serum glucose, lipid profile and serum biomarkers for plaque initiation (Lipid profile, LpPLA2), endothelial activation (MCP-1), plaque inflammation (hsCRP, IL6, IL18, TNF, advanced glycation end-products), vulnerable transformation (vEGF, PAI-1, BMP-6) and measures of oxidative stress (Ox-LDL, TAOS, TBARs) at baseline, and at 12 months after therapy initiation

SUMMARY:
Individuals with T2DM have a two-fold excess risk of cardiovascular (CV) events compared with their non-diabetic counterparts.

Although it is the primary cause of death in T2DM, there is no significant evidence that intensive glucose lowering reduces CV events. Multiple Cardiovascular Outcome Trials have suggested CV safety and benefit with the new class hypoglycemic agents - glucagon-like peptide 1 receptor agonists (GLP-RAs) in patients with DM and a high CV risk profile with a mechanism not directly dependent on their glucose-lowering effect. Varies theories regarding the mechanism of action of GLP-RAs on reducing CV events have been proposed, including reducing inflammation, protection of ischemia/reperfusion injury, and improvement in endothelial dysfunction but the effects of these new agents on in-vivo atherosclerotic plaque burden is currently unproven.

The investigators hypothesize that compared with placebo, 1-year treatment with the oral GLP-RA "Semaglutide" will result in a regression of necrotic core within potentially vulnerable coronary plaques (identified using the novel method "Plaque Maps" analysis on CT Coronary Angiography) in patients with raised HbA1c (>5.7%) after acute coronary syndromes (ACS).

Methods: One hundred forty patients admitted with ACS and have raised HbA1c >5.7% will be enrolled in the trial and randomized in a 1:1 blinded fashion to receive conventional therapy and initiation of Semaglutide or conventional therapy plus placebo.

All patients will have a CT Coronary Angiography with Plaque Map analysis of atherosclerotic burden, plaque composition and presence of potentially vulnerable plaque morphology at baseline prior to therapy initiation and following 12 months of treatment. In addition, to help elucidate the potential mechanisms of any anti-atherosclerotic effects, patients will have a non-invasive assessment of vascular function assessed by aortic pulse wave velocity and comprehensive biomarker analysis of inflammation, atherogenesis and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c > 5.7% (39 mmol/mol)
* Patients presented with a clinical diagnosis of ACS comprising detection of a rise and/or fall of cardiac troponin (cTn) with at least one value above the 99th percentile and with at least one of the following:

  1. Symptoms of acute myocardial ischemia;
  2. New ischemic electrocardiographic (ECG) changes (ST-T wave changes or new LBBB);
  3. Development of pathological Q waves;
  4. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischemic aetiology;
  5. Identification of a coronary thrombus by angiography including intracoronary imaging or by autopsy

Exclusion Criteria:

* Type 1 DM
* Left ventricular ejection fraction <40%
* Heart failure classified as being in New York Heart Association (NYHA) Class III-IV.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within the past 90 days prior to screening or in the period between screening and randomisation.
* History of renal insufficiency with estimated glomerular filtration rate <30mL/min/1.73m2
* A personal or family history of medullary thyroid carcinoma (MTC) or in patients with Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* History of treatment with GLP-1 within 90 days before screening
* Current use of SGLT-2 inhibitors within 30 days of screening
* Known or suspected hypersensitivity to Semaglutide or related products.
* Female who is pregnant, breastfeeding or intends to become pregnant, or is of child-bearing potential and not using a highly effective contraceptive method.
* Current enrolment in any other clinical trial within 30 days from screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Compare the regression of vulnerable coronary plaque (necrotic core) assessed using histologically validated "Plaque Maps" derived from CT Coronary angiography in patients with raised HbA1c admitted with ACS and treated with oral Semaglutide or placebo. | 12 months
  Reduction in mean coronary plaque necrotic core (%) identified by CT Coronary Angiography Plaque Maps after 12-month therapy (Semaglutide or placebo).

SECONDARY OUTCOMES:
-Evaluate the effect of oral Semaglutide on atherosclerotic plaque burden. | 12 months
  Compare the regression (or progression) of vulnerable coronary plaque burden (%) assessed by CTCA in patients treated with oral Semaglutide or placebo for 12 months.
Evaluate the effect of oral Semaglutide on levels of biomarkers of inflammation. | 12 months
  Assess the changes in levels of serum biomarkers for inflammation (inflammation (hsCRP, IL6, IL18, TNF, advanced glycation end-products) at baseline, and at 12 months after therapy initiation (Drug vs placebo).
  The biomarkers will be calculated on the whole as one outcome. i.e. if the majority of the biomarkers are decreasing with the use of oral Semaglutide , this will count as a positive outcome and vice versa.
  Every biomarker value will be recorded in the trial before and after the follow-up period
-Evaluate any potential effect of oral Semaglutide on arterial stiffness | 12 months
  Assess the changes in arterial stiffness by calculating aortic carotid-femoral pulse wave velocity (cfPWV) through the Vicorder (Skidmore medical, UK) at baseline, and at 12 months after therapy initiation (Drug vs placebo).
Evaluate the effect of oral Semaglutide on levels of biomarkers of oxidative stress. | 12 months
  Assess the changes in levels of serum biomarkers for oxidative stress (Ox-LDL, TAOS, TBARs) at baseline, and at 12 months after therapy initiation (Drug vs placebo).
  The biomarkers will be calculated on the whole as one outcome. i.e. if the majority of the biomarkers are decreasing with the use of oral Semaglutide , this will count as a positive outcome and vice versa.
  Every biomarker value will be recorded in the trial before and after the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Swansea Bay University Health Board, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No